CLINICAL TRIAL: NCT05149729
Title: Mid-Term Natural Course of Lower Extremity and Spine After Total Hip Arthroplasty in Patients With Crowe Type III-IV Hip Dysplasia
Brief Title: Mid-Term Natural Course Postoperative of Crowe Type III-IV Hip Dysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Murat Sarikas, Orthopaedic surgeon, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E.16313
Record Dates: First submitted 2021-10-08; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Hip Arthropathy; Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Intervention Model Description: Patients over the age of 18 who underwent Crowe Type 3 and Type 4 shortened hip prosthesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crowe type 3 and 4 patients undergoing shortened hip replacement (Experimental): Clinical and radiological results of Crowe type 3 and 4 patients who underwent shortened hip prosthesis at 12 and 24 months
  Interventions: Procedure: Shortened hip arthroplasty

INTERVENTIONS:
Procedure: Shortened hip arthroplasty — Crowe type 3 and 4 patients who underwent shortened hip prosthesis

SUMMARY:
Comparison of preoperative and postoperative mid-term course of patients with Crowe Type 3 and Type 4 hip dysplasia.

DETAILED DESCRIPTION:
Crowe type 3 and type 4 patients who underwent shortened hip replacement surgery will be followed up for 2 years.

Patients will be called for routine outpatient controls at the 2nd week, 6th week, 3rd month, 6th month, 12th month, 24th month.

Patients will be referred to the physical therapy specialist for abduction strengthening and pelvis tilt corrective exercises starting from the 6th week.

Scoliosis and orthoroentgenography x-rays will be taken at the last control of the patients.

HHS, WOMAC hip score and SF-12 score will be obtained from the patients. Scores, lower extremity and spine angles will be evaluated after the last examinations performed at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Crowe type 3 and 4 patients over 18 years of age who had shortened hip replacement surgery

Exclusion Criteria:

* Crowe type 1 or 2 patients over 18 years of age who had shortened hip replacement surgery
* Patients who have previously operated on the contralateral hip
* Patients who underwent shortened hip replacement for a reason other than developmental dysplasia of the hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | The degree of improvement in Vomac score will be evaluated by looking at preoperative and postoperative 12th month Vomac scores.( 0-12th month )
  The WOMAC score range, which indicates the clinical satisfaction of the patients, is between 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Gökçer Uzer, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EFFECTS OF TOTAL HIP ARTHROPLASTY ON AXIAL ALIGNMENT — https://DOI.ORG/10.1016/J.ARTH.2019.04.028
- See also: CHANGES IN HIP, KNEE, AND ANKLE CORONAL ALIGNMENTS AFTER TOTAL HIP ARTHROPLASTY WITH TRANSVERSE FEMORAL SHORTENING OSTEOTOMY FOR UNILATERAL CROWE TYPE IV DEVELOPMENTAL DYSPLASIA OF THE HIP — https://DOI.ORG/10.1016/J.ARTH.2017.05.044